CLINICAL TRIAL: NCT03670706
Title: The East-Midlands Knee Pain Multiple Randomised Controlled Trial Cohort Study: Cohort Establishment and Feasibility Cohort-randomised Controlled Trial
Brief Title: Knee Pain Nurse Led Package of CareTrial
Acronym: Team-KP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nottingham (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: Team-KP
Record Dates: First submitted 2018-09-04; First posted 2018-09-13 (Actual); Last update posted 2021-09-21 (Actual); Status verified 2021-09

CONDITIONS: Osteoarthritis, Knee; Pain, Joint
MeSH Terms: conditions — Osteoarthritis, Knee; Arthralgia | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (Active Comparator): Exercise training, then crossover to analgesic optimisation
  Interventions: Behavioral: Exercise; Other: analgesic optimisation
- Group B (Active Comparator): Analgesic optimisation, then crossover to exercise training
  Interventions: Behavioral: Exercise; Other: analgesic optimisation
- Group C (No Intervention): Control group

INTERVENTIONS:
Behavioral: Exercise — Package of care
  Other Names: Package of care
  Arms: Group A; Group B
Other: analgesic optimisation — optimisation
  Arms: Group A; Group B

SUMMARY:
1. To develop a training package for nurse-led management of knee osteoarthritis (OA), incorporating information about OA and core non-pharmacologic and pharmacologic principles of management of OA as recommended in the National Institute for Clinical Excellence and Health (NICE) guidelines for management of OA
2. To evaluate fidelity of delivery of individual components of this complex package of care for knee pain
3. To assess the acceptability of the intervention by exploring participant satisfaction with nurse-led complex package of care of knee pain.
4. To explore and resolve possible challenges to delivery of individual components within a complex package
5. To examine the feasibility of a definitive cohort randomised controlled trial of nurse-led care versus usual care of knee pain in terms of recruitment rate, drop-out rate, reasons for dropping out and completeness of outcome data
6. To explore whether such a trial should provide analgesia before non-pharmacologic interventions or vice versa

ELIGIBILITY:
Inclusion Criteria:

* Knee pain on most days of the previous month
* At least moderate pain on two of the five WOMAC knee pain domains in the most painful knee
* Knee pain present for longer than 3 months

Exclusion Criteria:• House-bound or care home resident

* Dementia
* Dialysis
* On home oxygen
* Serious mental illness
* Inability to communicate in English
* Unable to give consent
* Terminal cancer
* Known diagnosis of autoimmune rheumatic diseases or psoriasis
* Knee or hip replacement, or on waiting list for knee or hip replacement
* Asthma or COPD requiring regular daily oral corticosteroids
* Unstable angina or heart failure
* Known peripheral vascular disease
* Pregnant

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1806 (Actual)
Dates: Start 2018-11-26 (Actual); Primary Completion 2021-07-05 (Actual); Study Completion 2021-07-05 (Actual)

PRIMARY OUTCOMES:
The Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) | 26 weeks
  questionnairehe Western Ontario and McMaster Universities Arthritis Index (WOMAC) is widely used in the evaluation of Hip and Knee Osteoarthritis. It is a self-administered questionnaire consisting of 24 items divided into 3 subscales:
  Pain (5 items): during walking, using stairs, in bed, sitting or lying, and standing upright Stiffness (2 items): after first waking and later in the day Physical Function (17 items): using stairs, rising from sitting, standing, bending, walking, getting in / out of a car, shopping, putting on / taking off socks, rising from bed, lying in bed, getting in / out of bath, sitting, getting on / off toilet, heavy domestic duties, light domestic duties

CONTACTS AND LOCATIONS:
Overall Officials: Abhishek Abhishek, Principal Investigator — University of Nottingham/ Nottingham University NHS Trust
Locations (1):
- Nottingham University Hospitals NHS Trust, Nottingham, United Kingdom

REFERENCES:
- [Derived] Fuller A, Hall M, Nomikos PA, Millar B, Ogollah R, Valdes A, Greenhaff P, das Nair R, Doherty M, Walsh DA, Abhishek A. Feasibility of conducting a cohort randomized controlled trial assessing the effectiveness of a nurse-led package of care for knee pain. Rheumatology (Oxford). 2024 May 3;63(6):1582-1592. doi: 10.1093/rheumatology/kead432. PMID 37610332
- [Derived] Nomikos PA, Hall M, Fuller A, Millar B, Ogollah R, Valdes A, Doherty M, Walsh DA, das Nair R, Abhishek A. Fidelity assessment of nurse-led non-pharmacological package of care for knee pain in the package development phase of a feasibility randomised controlled trial based in secondary care: a mixed methods study. BMJ Open. 2021 Jul 29;11(7):e045242. doi: 10.1136/bmjopen-2020-045242. PMID 34326044
- [Derived] Hall M, Fuller A, Nomikos PA, Millar B, Ogollah R, Valdes A, Greenhaff P, das Nair R, Doherty M, Walsh DA, Abhishek A. East Midlands knee pain multiple randomised controlled trial cohort study: cohort establishment and feasibility study protocol. BMJ Open. 2020 Sep 9;10(9):e037760. doi: 10.1136/bmjopen-2020-037760. PMID 32912951